CLINICAL TRIAL: NCT00251888
Title: Etude de Recherche de Dose de l'Association Irinotecan (Campto(R)) - Cisplatine (Cisplatyl(R)) Avec la radiothérapie Pelvienne Dans Les Cancers avancés du Col de l'utérus.
Brief Title: CAmpto-CISplatine Plus Radiotherapy in Advanced Cervix Cancer : Search of Tolerated Maximum Dose of Campto
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: ARCAGY/ GINECO GROUP (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CACIS
Record Dates: First submitted 2005-11-10; First posted 2005-11-11 (Estimated); Last update posted 2017-01-25 (Estimated); Status verified 2011-02

CONDITIONS: Cervix Cancer
Keywords: cervix cancer; advanced cervix cancer; radiochemotherapy; pelvic radiotherapy; campto; cisplatin; irinotecan; cisplatyl; maximum dose search
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Irinotecan; Cisplatin

INTERVENTIONS:
Drug: campto (irinotecan)
Drug: cisplatin (cisplatyl)

SUMMARY:
Search of maximum tolerated irinotecan dose in association with cisplatin and pelvic radiotherapy in patients with an advanced cervix cancer.

DETAILED DESCRIPTION:
To determine the maximum and the recommended tolerated dose of irinotecan with increasing doses associated with weekly cisplatin and combinated with pelvic radiotherapy in patients with an advanced cervix cancer, IIB-IVA FIGO stage.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven primitive epidermoid or andenocarcinoma Cervix
* FIGO stage IIB (obviously parameter attack), III or IVA
* No previous chemotherapy nor radiotherapy
* Patient for whom a radiochemotherapy is envisaged as first intention treatmentof her cervix carcinoma
* PS ECOG < 2
* Life expectancy > 12 weeks
* Written consent given

Exclusion Criteria:

* Other malignant cervix tumor histology
* Visceral remotly metastasis
* Other malignant tumor since 5 years, except spino or baso-cellular treaten and cured cancer
* Anormal labs values
* Peripheric neuropathy CTC > 2
* Auditory loss > 2
* Cardiopathy
* Inflammatory digestive pathology
* Evolutive infection
* Other experimental concommitant treatment
* Lacting or pregnant women

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15
Dates: Start 2002-11; Study Completion 2005-11 (Actual)

PRIMARY OUTCOMES:
To determine the maximum tolerated dose of irinotecan associated with cisplatin and combinated with pelvic radiotherapy in patients with an advanced cervix cancer

SECONDARY OUTCOMES:
To evaluate :
the global response rate judged on standard clinical criteria, echography, tomodensiometry, and MRI. The histologic response rate will be appreciated in patients who had a second surgery after pelvic radiochemotherapy
local and general relapse frequency
progression free survival
global survival

CONTACTS AND LOCATIONS:
Overall Officials: Christophe Hennequin, Physician, Principal Investigator — Hôpital St Louis, Paris, France; Nadine Dohollou, physician, Principal Investigator — Clinique Bordeaux Nord, Bordeaux, France
Locations (2):
- France (2):
  - CRLC Val d'Aurelle, Montpellier
  - Centre Claudius Régaud, Toulouse